CLINICAL TRIAL: NCT06299553
Title: INCB88888-040 Multicenter Prospective Real-world Observational Cohort Study to Evaluate the Effectiveness of Tafasitamab in Combination With Lenalidomide Followed by Tafasitamab Monotherapy in Relapsed or Refractory Diffuse Large B-cell Lymphoma Non-transplant Eligible Patients in Italy (PRO-MIND)
Brief Title: Study to Evaluate the Effectiveness of Tafasitamab in Combination With Lenalidomide Followed by Tafasitamab Monotherapy in Relapsed or Refractory Diffuse Large B-cell Lymphoma Non-transplant Eligible Patients in Italy (PRO-MIND)
Status: Recruiting | Type: Observational
Sponsor: Incyte Biosciences Italy S.r.l (Industry)
Collaborators: Advice Pharma Group srl (Industry)
Responsible Party: Sponsor
Other Study IDs: INCB88888-040 PRO-MIND
Record Dates: First submitted 2024-02-22; First posted 2024-03-08 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma
Keywords: Tafasitamab; Lenalidomide
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group/cohort: Patients with DLBCL R/R disease non-transplant eligible

SUMMARY:
The PRO-MIND study is an Italian, multicenter, prospective observational cohort study to evaluate the effectiveness and the safety of tafasitamab in combination with lenalidomide followed by tafasitamab monotherapy in patient with DLBCL.

DETAILED DESCRIPTION:
This is an Italian, multicenter, prospective observational cohort study to collect data on patients with non-transplant eligible R/R DLBCL treated with tafasitamab plus lenalidomide followed by tafasitamab in monotherapy, as second, third and fourth treatment line in a real-world clinical practice setting.

The study is non-interventional; all treatment decisions are made at the discretion of the patient's healthcare provider and are not mandated by the study design or protocol.

Since this is an observational study of real-world treatment practices and outcomes, no study medication will be provided as a part of this study. Tafasitamab and lenalidomide will be provided through usual commercial channels for medicines prescription. Tafasitamab and lenalidomide will not be provided free of charge by the sponsor.

Physicians will make all treatment decisions according to their usual clinical practices and will provide prescriptions for their patients as appropriate. The decision to treat the patient with tafasitamab must have been taken prior to and independently of the patient's inclusion in the study. There are no mandatory protocol procedures or diagnostic tests.

This is a prospective observational study: patients will be eligible to enter the study if the treatment with tafasitmab plus lenalidomide is started and when all the ethical and contract procedures with the site have been completed and after the site initiation visit date.

The study will be performed in approximately 30 Italian sites distributed in the overall Italian territory.

During this study, patients must completed questionnaires of quality of life. Questionnaires should be completed by the patient Electronic Patient Reported Outcome (ePRO)at each applicable occasion. Where possible in accordance with local clinical practice, PROs should be completed before other assessments. The following measures are requested to be recorded:

* EORTC-QLQ-C30 (Version 3).
* EORTC QLQ NHL-HG29

The standardized EORTC QLQ-C30 questionnaire (v. 3.0) was used to assess the HRQoL of cancer patients. The questionnaire contains questions regarding the impact of the disease on different areas of a patient's life (physical, role, emotional, cognitive, and social functioning), the occurrence of symptoms (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, and diarrhea), financial difficulties, and an overall assessment of HRQoL (Appendix 4). (Aaronson NK, Ahmedzai S, Bergman B, et al. 1993). For each question, the respondent must choose 1 answer. For 28 of the questions, the answers are given on a 4-point Likert-type scale (1 - never, 2 - sometimes, 3 - often, 4 - very often) and assess the intensity of the analysed parameters. The last 2 questions evaluate the general health of the patient on a 7-point scale (from 1 - very bad to 7 - excellent). Patients completed the questionnaires by themselves. If a question arose, they could ask the researcher for an explanation.

After collecting the responses, a raw score was calculated for each of the abovementioned 15 questionnaire items. Next, a linear transformation was performed to obtain a score in a range from 0 to 100. The conversion of the results to a 100-point scale was made according to the EORTC guidelines. Of note, a higher score on the functional scales means better functioning and a higher response for general health corresponds to a better HRQoL.

The QLQ-HG-NHL29 consists of 29 items, contributing to five multiitem subscales and three conditional items: symptom burden due to disease and/or treatment (seven items), neuropathy (two items), physical condition/fatigue (five items), emotional impacts (four items) and worries about health and functioning (eight items). The three conditional items, which patients complete only if relevant to them, are about having problems at work/education, worries about work/education and concerns about the ability to have children. (Appendix 5) (Van de Poll-Franse L, Oerlemans S, Bredart A, et al. 2018) Items are rated using a four-point response scale ("not at all," "a little," "quite a bit," and "very much") and the reference time frame for all items is the past week.14 The scoring approach for the QLQ-HG-NHL29 is identical to that of the EORTC QLQ-C30, i.e., calculating the mean of the items of a specific multi-item scale or using the single conditional item score and then converting it into a standardized scale ranging from 0 to 100. A higher score for all the multi-item scales and items represent a higher level of symptomatology or problems.

HRQoL questionnaires will be filled out either at the hospital or during pre-scheduled medical office visits. The questionnaires will be provided to the patient by a member of the study team at the scheduled times to coincide with other scheduled assessments or visits, via standard paper copy administration. However, HRQoL electronic questionnaires administration may be allowed as a back-up procedure, to maximize compliance. Patients will be asked to fill out the questionnaires as completely and accurately as possible with an expected average time of completion around 10 minutes.

A high compliance with HRQoL questionnaires throughout the study period is considered essential for the success of this observational study and local Investigators of participating centers will have to be properly informed and motivated towards the importance of collecting HRQoL data.

Each participating center will be requested to submit a HRQoL Missing Data Form in lieu of a HRQoL questionnaire for any assessment that is not provided at the appropriate follow-up time point. Compliance with HRQoL questionnaires over time will be monitored (not for the purpose of informing clinical care of participants) and, if needed, reminders will be sent to participating centers to solicit HRQoL data. The compliance rate at each time point will be evaluated as the number of valid HRQoL questionnaires returned by eligible patients as a proportion of the total number of eligible patients available.

In order to make the HRQoL component of the study as pragmatic as possible, and not to undermine the data collection process across several centers, HRQoL assessment is requested to take place in conjunction with the collection of effectiveness data foreseen for this protocol.

Therefore, HRQoL questionnaires will be administered at baseline (before first tafasitamab administration) and then every 3 months during the first year, and then every 6 months thereafter, unless the patient has a disease progression and/or permanently discontinue treatment with tafasitamab. The first HRQoL assessment after baseline, would correspond to the end of the period where tafasitamab is administered on a weekly basis (approximately at the end of cycle 3), hence with potential expected HRQoL detriments. Thereafter, (starting from cycle 4) considering the infusions of tafasitamab will take place every 2 weeks, HRQoL improvements (although with not known magnitude) could possibly be expected and captured in this study. HRQoL will be assessed regardless of dose modification or temporary treatment interruption, as long as the patient is considered "on study" according current protocol definition.

In case of temporary treatment interruption:

Continue HRQoL assessment as described in the above schedule of administration.

In case of permanent treatment discontinuation with tafasitamab:

HRQoL assessment should be performed at the time of discontinuation (in any case as close as possible to the time of treatment discontinuation) and then stopped afterwards.

In case of disease progression:

HRQoL assessment should be performed at the time of progression (in any case as close as possible to the time of disease progression) and then stopped afterwards.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are aged 18 years or older.
2. Patients with DLBCL R/R disease non-transplant eligible.
3. Patients who will initiate the treatment with commercially available tafasitamab and lenalidomide after the ICF signature. The decision to prescribe tafasitamab must have been made prior and regardless of the enrollment of the patient in the study.
4. Patients are able of giving the signed informed consent.

Exclusion Criteria:

1. Concomitant participation in an interventional clinical study
2. Any patient in the physician's opinion from whom initial diagnosis or follow-up data is unlikely to be obtained reliably data for the purposes of this observational study.
3. Patients who started tafasitamab treatment before signing the ICF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The enrollment will be done consecutively and starting from the list of patients identified in the Screening/Enrollment Log. Participating sites will be encouraged to enroll patients in a consecutive manner when patients come for their regular visit, in order to minimize bias in patient selection. At each participating site, the physician will assess patients to determine their eligibility for data collection within the study based on the selection criteria listed below. All patients will give their informed consent to participate in this study and will sign privacy disclosure before data collection is performed. All subjects documented are being treated according to local labeling specifications.The inclusion/exclusion criteria reflect the current approved Summary of Product Characteristics (SmPC) and AIFA monitoring registry.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | At the beginning of Cycle 1 (day 1 of this cycle. The duration of each cycle is 28 days), visit in the 1° year (every 3 months) and visit in the 2°, 3°, 4° years (every 6 months).
  PFS is defined as the time from the date of treatment initiation until the first documented progression or relapse of disease measured by routine clinical care by the physician.

SECONDARY OUTCOMES:
Baseline Characteristics | Baseline, At the beginning of Cycle 1 (day 1 of this cycle. The duration of each cycle is 28 days), visit in the 1° year(every 3 months) and visit in the 2°, 3°, 4° years(every 6 months).
  Demographics and clinical characteristics of patients receiving tafasitamab
Overall Response Rate (ORR) | Visit in the 1° year (every 3 months) and visit in the 2°, 3°, 4° years (every 6 months).
  Percentage of patients who have met the ORR definition up until progression based on the physician's assessment.
Duration of Response (DoR) | Visit in the 1° year (every 3 months) and visit in the 2°, 3°, 4° years (every 6 months).
  The time interval between the initial time point of tumor response (CR or PR whichever status is recorded first) and the first date that recurrence of progressive disease is documented as physician assessment.
Time to next treatment (TTNT) | At the beginning of Cycle 1 (day 1 of this cycle. The duration of each cycle is 28 days), visit in the 1° year (every 3 months) and visit in the 2°, 3°, 4° years (every 6 months).
  The time from first tafasitamab dosing to the institution of next therapy for any reason including disease progression, treatment toxicity and patient preference.
Time to response | Visit in the 1° year(every 3 months) and visit in the 2°, 3°, 4° years (every 6 months).
  To determine the time to response, defined as the time from first tafasitamab dosing to the first response (each response or CR).
Overall Survival (OS) | Cycle 1 day 1, Visit in the 1° year(every 3 months) and visit in the 2°, 3°, 4° years (every 6 months).
  OS defined as the time from the date of treatment initiation until death from any cause
Disease Control Rate (DCR) | Baseline, At the beginning of Cycle 1 (day 1 of this cycle. The duration of each cycle is 28 days), Visit in the 1° year (every 3 months) and visit in the 2°, 3°, 4° years (every 6 months)
  Percentage of patients who have met the DCR definition during treatment based on the physician's assessment.
Event Free Survival (EFS) | Visit in the 1° year(every 3 months) and visit in the 2°, 3°, 4° years (every 6 months).
  The time from first tafasitamab dose to an event which may include disease progression, discontinuation of the treatment for any reason, or death.
Progression-Free-Survival 2 (PFS2) | Visit in the 1° year (every 3 months) and visit in the 2°, 3°, 4° years (every 6 months).
  The time from first tafasitamab dose to progression on first subsequent therapy as per physician assessment.
Information of which treatment the patients will get after tafasitamab discontinuation | Visit in the 1° year (every 3 months) and visit in the 2°, 3°, 4° years (every 6 months)
  Name of the treatment after tafasitamab discontinuation.
Safety of tafasitamab combined with lenalidomide | At the beginning of Cycle 1 (day 1 of this cycle. The duration of each cycle is 28 days), Visit in the 1° year (every 3 months) and visit in the 2°, 3°, 4° years (every 6 months)
  Percentage of patients with serious and non-serious adverse events (AEs/ADRs/SAEs and SADRs) treated with tafasitamab plus lenalidomide.
Safety of tafasitamab in monotherapy | At the beginning of Cycle 1 (day 1 of this cycle. The duration of each cycle is 28 days), Visit in the 1° year(every 3 months) and visit in the 2°, 3°, 4° years (every 6 months)
  Percentage of patients with serious and nonserious adverse events (AEs/ADRs/SAEs and SADRs) treated with tafasitamab alone.
Describe the treatment adherence of lenalidomide and dose reduction. | At the beginning of Cycle 1 (day 1 of this cycle. The duration of each cycle is 28 days), Visit in the 1° year (every 3 months) and visit in the 2°, 3°, 4° years (every 6 months)
  Percentage of patients with Medical Possession Rate (MPR) >=80% and dosing.
Health-Related Quality of Life (HRQoL) | Baseline, Visit in the 1° year(every 3 months) and visit in the 2°, 3°, 4° years (every 6 months).
  The HRQoL consisted of 30 questions. 28 of the questions, the answers are given on a 4-point Likert-type scale (1 - never, 2 - sometimes, 3 - often, 4 - very often) and assess the intensity of the analysed parameters. The last 2 questions evaluate the general health of the patient on a 7-point scale (from 1 - very bad to 7 - excellent).
Health-Related Quality of Life (HRQoL) | Baseline, Visit in the 1° year(every 3 months) and visit in the 2°, 3°, 4° years (every 6 months).
  The QLQ-HG-NHL29 consists of 29 items, contributing to five multiitem subscales and three conditional items: symptom burden due to disease and/or treatment (seven items), neuropathy (two items), physical condition/fatigue (five items), emotional impacts (four items) and worries about health and functioning (eight items). The three conditional items, which patients complete only if relevant to them, are about having problems at work/education, worries about work/education and concerns about the ability to have children. Items are rated using a four-point response scale ("not at all," "a little," "quite a bit," and "very much") and the reference time frame for all items is the past week.
Health economics - Hospitalization | Visit in the 1° year (every 3 months) and visit in the 2°, 3°, 4° years (every 6 months)
  Duration of hospitalization (total days length of stay, including duration by wards, eg, intensive care unit)
Health economics - DLBCL treatment | Visit in the 1° year (every 3 months) and visit in the 2°, 3°, 4° years (every 6 months)
  Treatments administered during the hospitalization
  * To explore possible factors associated with the effectiveness of tafasitamab (prediction of response);
  * To describe the CD19 expression status before and after the tafasitamab treatment, if done in clinical practice.
Health economics - Concomitant Treatments | Visit in the 1° year (every 3 months) and visit in the 2°, 3°, 4° years (every 6 months)
  Concomitant treatments (i.e. supportive treatments) administered to the patient (dosage, number of administrations, way of administration)
Health economics - Monitoring activities | Visit in the 1° year (every 3 months) and visit in the 2°, 3°, 4° years (every 6 months)
  Monitoring activities performed during the hospitalization (i.e. laboratory tests, imaging procedures, visits)
Health economics - monitoring activities performed after patients' discharge | Visit in the 1° year (every 3 months) and visit in the 2°, 3°, 4° years (every 6 months)
  Monitoring activities performed after patient's discharge (i.e. laboratory tests, imaging procedures, visits)
Health economics - Adverse event treatment | Visit in the 1° year (every 3 months) and visit in the 2°, 3°, 4° years (every 6 months)
  Adverse events treatment: per each adverse event, the activities performed to manage it will be assessed in terms of laboratory tests (type and number), imaging procedures (type and number), drugs (dosage, number of administrations, way of administration), visits, medical procedures (type and number)
Health economics - Unplanned specialist visits | Visit in the 1° year (every 3 months) and visit in the 2°, 3°, 4° years (every 6 months)
  Unplanned specialist visits that occurred between FU visits
Exploratory objectives | Baseline, At the beginning of Cycle 1 (day 1 of this cycle. The duration of each cycle is 28 days), Visit in the 1° year (every 3 months) and visit in the 2°, 3°, 4° years (every 6 months)
  possible factors associated with the effectiveness of tafasitamab (prediction of response)
Exploratory objectives | Baseline, At the beginning of Cycle 1 (day 1 of this cycle. The duration of each cycle is 28 days), Visit in the 1° year (every 3 months) and visit in the 2°, 3°, 4° years (every 6 months)
  CD19 expression status before and after the tafasitamab treatment, if done in clinical practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Incyte Biosciences Italy S.r.l, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zinzani PL, Minotti G. Anti-CD19 monoclonal antibodies for the treatment of relapsed or refractory B-cell malignancies: a narrative review with focus on diffuse large B-cell lymphoma. J Cancer Res Clin Oncol. 2022 Jan;148(1):177-190. doi: 10.1007/s00432-021-03833-x. Epub 2021 Nov 6. PMID 34741682
- [Background] Duell, J., Abrisqueta, P., Andre, M., Augustin, M., Gaidano, G., Barca, E.G., Jurczak, W., Kalakonda, N., Liberati, A.M., Maddocks, K.J., Menne, T., Nagy, Z., Tournilhac, O., Bakuli, A., Amin, A., Gurbanov, K. and Salles, G. (2023), Five-year efficacy and safety of tafasitamab in patients with relapsed or refractory DLBCL: Final results from the Phase II L-MIND study. Hematological Oncology, 41: 437-439
- [Background] Calamia M, McBride A, Abraham I. Economic evaluation of polatuzumab-bendamustine-rituximab vs. tafasitamab-lenalidomide in transplant-ineligible R/R DLBCL. J Med Econ. 2021 Nov;24(sup1):14-24. doi: 10.1080/13696998.2021.2007704. PMID 34866523
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] van de Poll-Franse L, Oerlemans S, Bredart A, Kyriakou C, Sztankay M, Pallua S, Daniels L, Creutzberg CL, Cocks K, Malak S, Caocci G, Molica S, Chie W, Efficace F; EORTC Quality of Life Group. International development of four EORTC disease-specific quality of life questionnaires for patients with Hodgkin lymphoma, high- and low-grade non-Hodgkin lymphoma and chronic lymphocytic leukaemia. Qual Life Res. 2018 Feb;27(2):333-345. doi: 10.1007/s11136-017-1718-y. Epub 2017 Nov 10. PMID 29127596